CLINICAL TRIAL: NCT01711957
Title: The Perioperative Value of Platelet Counts in Predicting Outcome After Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Dimitri Aristotle Raptis, MD, PhD, University of Zurich
Other Study IDs: EK-1487
Record Dates: First submitted 2012-10-18; First posted 2012-10-23 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Complication; Death
Keywords: Complications; Mortality; Liver transplantation; Platelet count; Survival
MeSH Terms: conditions — Death | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liver disease and liver transplantation: Patient with end stage liver disease and/or primary liver tumor undergoing liver transplantation
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Standardized technique of liver transplantation Organ procurement follow the rules of the Swiss transplant society
  Other Names: Orthotopic liver transplantation (OLT); Cadaveric-donor liver transplantation

SUMMARY:
Recent experimental and clinical studies have shown that platelets play a critical role in liver ischemia and regeneration. Thrombocytopenia, a frequent and potentially serious condition in liver transplantation (LT) recipients, was shown to be associated with postoperative morbidity and mortality after partial hepatectomy.

The investigators aim at evaluating whether postoperative low platelet counts are indicators of short- and long-term outcomes after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* End stage liver disease
* Cadaveric-donor liver transplantation

Exclusion Criteria:

* Age <18 years old
* Pregnancy
* Living-related liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end stage liver disease and/or primary liver tumor undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Severe complication after liver transplantation | 90 days
  The severity of complications will be graded according to the Clavien-Dindo classification by outcome. Grade III to V complications will be considered as severe.

SECONDARY OUTCOMES:
Primary graft non-function | first postoperative week
  Defined as death or retransplantation within the first postoperative week after exclusion of technical, immunological, and infectious causes
Delayed graft function | 7 days after liver transplantation
  Defined as the presence of at least one of the following parameter at 7 days after LT: serum bilirubin > 10 mg/dL and International Normalized Ratio (INR) >1.6 or Alanine aminotransferase serum level (ALT) >2000UI/L

OTHER OUTCOMES:
Patient survival | 3-year

CONTACTS AND LOCATIONS:
Overall Officials: Mickael Lesurtel, M.D., PhD, Study Director — University of Zurich; Pierre-Alain Clavien, M.D., PhD, Study Chair — University of Zurich; Dimitri A. Raptis, M.D., MSc, Principal Investigator — University of Zurich; Emmanuel Melloul, M.D., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Department of Visceral Surgery and Transplantation, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Lesurtel M, Raptis DA, Melloul E, Schlegel A, Oberkofler C, El-Badry AM, Weber A, Mueller N, Dutkowski P, Clavien PA. Low platelet counts after liver transplantation predict early posttransplant survival: the 60-5 criterion. Liver Transpl. 2014 Feb;20(2):147-55. doi: 10.1002/lt.23759. Epub 2013 Nov 21. PMID 24123804